CLINICAL TRIAL: NCT00353548
Title: Study of Response to the Taste of Beverages That Are Not Swallowed (Sipping and Spitting in Eating Disorders)
Brief Title: Determining the Response to Sipping Beverages Without Swallowing in People With Eating Disorders
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5046/#6158R; K23MH071285-01 (NIH); DATR AK-TNAI1
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Eating Disorders
Keywords: Bulimia Nervosa; Binge Eating Disorder; Obesity; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder; Obesity; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1-Anorexia Nervosa: Women ages 16-50 who meet DSM-IV criteria for anorexia nervosa
- 2-Bulimia Nervosa: Women age 16-50 who meet DSM-IV criteria for bulimia nervosa
- 3-Binge Eating Disorder: Women with binge eating disorder
- 4-Healthy Controls: Healthy control subjects ages 16-50 of normal weight
- 5-Obese Controls: Healthy obese control subjects

SUMMARY:
This study will use a sipping and spitting exercise to better understand the brain's response to food intake in people with eating disorders.

DETAILED DESCRIPTION:
Eating behavior is controlled by many factors, including appetite; food availability; family, peer, and cultural practices; and attempts at voluntary control. Eating disorders are characterized by a voluntary control of eating behavior, causing serious disturbances in normal eating habits. People with eating disorders demonstrate an extreme and unhealthy reduction or increase in food intake, as well as feelings of distress or extreme concern about body shape or weight. The three most common types of eating disorders are anorexia nervosa, bulimia nervosa, and binge eating disorder. People with anorexia nervosa have an intense fear of gaining weight or becoming fat. They are usually underweight, and resist maintaining a body weight at or above the minimum normal weight for their age and height. People with bulimia nervosa are less frequently underweight. Their eating habits are characterized by episodes of bingeing, followed by episodes of purging. Similarly, people with binge eating disorder have eating habits characterized by episodes of binge eating, but no purging. Studies on the basic biology of appetite control and the effects of overeating and starvation have revealed extensive information about eating disorders, but there are still questions to be answered. This study will use a sipping and spitting exercise to better understand the brain's response to food intake in people with eating disorders.

Participants in this observational study will first report to the Biological Studies Unit (BSU) for a screening visit. Participants will be provided with a series of sweetened beverages to taste and spit out. The beverages will be made with water, Kool-Aid mix, and sugar or artificial sweetener. Participants will rate the sweetness of each beverage and how much they like it. They will then practice sipping the beverage through a straw and spitting it out without swallowing. Those participants who feel comfortable with the sipping and spitting exercise will report to the BSU for 10 sipping and spitting exercises. The exercises may be scheduled on up to 4 separate days, and may last up to 2 hours per day. Participants will eat a standardized breakfast on the morning of the study, and then will not eat again until they report to the BSU 4 hours later. Participants will sit alone in a room alone, and sip and spit beverages for up to 5 minutes at a time. Between sipping and spitting sessions, participants will complete surveys about hunger and other sensations. They will also rinse their mouths out with baking soda and water to clear the taste of the previous beverage and to prevent discoloration of the mouth from the Kool-Aid. Measurements will include the amount of beverage sipped at a time, and how quickly each was sipped.

ELIGIBILITY:
Inclusion Criteria:

For participants with bulimia nervosa:

* Meets DSM-IV criteria for bulimia nervosa
* Duration of illness is 1 year
* Self-induces vomiting
* Weighs between 85 and 120% of ideal weight

For participants with anorexia nervosa:

* Meets DSM-IV criteria for anorexia nervosa (amenorrhea will not be required for study inclusion)
* Medically stable

For participants with binge eating disorder:

* Meets DSM-IV criteria for binge eating disorder
* Duration of illness is 1 year
* Body Mass Index (BMI) is at least 30

For healthy participants:

* Weighs between 80 and 120% of ideal weight

Exclusion Criteria:

For participants with anorexia nervosa, bulimia nervosa, or binge eating disorder:

* Significant medical illness
* At risk for suicide
* Currently taking medication
* History of drug or alcohol abuse within 6 months prior to study entry
* Pregnant or breastfeeding
* Axis I psychiatric disorder requiring pharmacotherapy
* Axis I psychiatric disorder that could impair ability to participate in the study (e.g., mania, psychosis)
* Comorbid binge eating disorder and an Axis I illness other than major depression

For healthy participants:

* Current or history of psychiatric illness
* History of any eating disorder
* Significant medical illness
* Currently taking medication
* History of drug or alcohol abuse within 6 months prior to study entry
* Pregnant or breastfeeding

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with anorexia nervosa, bulimia nervosa, and binge eating disorder as well as gender, age, and weight-matched control participants.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane A. Klein, MD, Principal Investigator — Columbia University Department of Psychiatry/New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States